CLINICAL TRIAL: NCT02828657
Title: ORBERA™ Post-Approval Study
Acronym: OPAS-1
Status: Completed | Type: Observational
Sponsor: Apollo Endosurgery, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OPAS-1
Record Dates: First submitted 2016-06-28; First posted 2016-07-11 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Obesity; Overweight
Keywords: ORBERA
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A prospective, multicenter, open-label, post-approval study of the safety and effectiveness of ORBERA™ as an adjunct to weight reduction for obese adults (22 years of age and older) with a Body Mass Index (BMI) of ≥ 30 kg/m2 and BMI ≤ 40 kg/m2

DETAILED DESCRIPTION:
FDA post-approval study designed to demonstrate the safety and effectiveness of ORBERA™ as an adjunct to weight reduction for obese adults (22 years of age and older) with a Body Mass Index (BMI) of ≥ 30 kg/m2 and BMI ≤ 40 kg/m2. Behavioral modification program in conjunction with endoscopic placement of a single ORBERA™ Intragastric Balloon, filled with saline to an inflation volume between 400cc and 700cc, for 26 weeks followed by endoscopic ORBERA™ removal. Outcomes include the mean percent Total Body Weight Loss (%TBWL), changes in weight, device and procedure-related AEs and SAEs: gastric ulcers, esophageal injury, placement and removal related SAEs, early device removals, and balloon deflations.

ELIGIBILITY:
Inclusion Criteria:

1. 22 years of age and older;
2. BMI ≥ 30 kg/m2 and ≤ 40 kg/m2;
3. Have a history of obesity (BMI ≥ 30 kg/m2) for ≥ 2 years;
4. Have failed more conservative weight-reduction alternatives, such as supervised diet, exercise, and behavioral modification programs;
5. Be willing to commit to a long-term supervised diet and behavior modification program designed to increase the possibility of long-term weight loss maintenance;
6. Be able to follow the requirements outlined in the protocol, including complying with the visit schedule;
7. Be able to provide written informed consent;

Exclusion Criteria:

1. Presence of more than one intragastric balloon at the same time;
2. Prior gastrointestinal surgery;
3. Has any inflammatory disease of the gastrointestinal (GI) tract including esophagitis, gastric ulceration, duodenal ulceration, cancer or specific inflammation such as Crohn's disease;
4. Has any gastrointestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasis, or other congenital anomalies of the GI tract such as atresias or stenosis;
5. Has a large hiatal hernia or hernia > 5 cm hernia or ≤ 5 cm associated with severe or intractable gastro-esophageal reflux symptoms;
6. Has a structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the delivery catheter and/or an endoscope;
7. Has achalasia or any other severe motility disorder that may pose a safety risk during removal of the device;
8. Has a gastric mass;
9. Has a severe coagulopathy;
10. Has hepatic insufficiency or cirrhosis;
11. Has any other medical condition which would not permit elective endoscopy, such as poor general health or history and/or symptoms of severe renal, hepatic, cardiac, and/or pulmonary disease;
12. Has serious or uncontrolled psychiatric illness or disorder that could compromise subject understanding of or compliance with follow-up visits and removal of the device after 6 months;
13. Alcoholism or drug addiction;
14. Unable or unwilling to take prescribed proton pump inhibitor medication for the duration of device placement;
15. Unwilling to participate in an established medically-supervised diet and behavior modification program, with routine medical follow-up;
16. Taking a daily dose of aspirin, anti-inflammatory agents, anticoagulants or other gastric irritants routinely and not under medical supervision;
17. Females who are pregnant, nursing, or planning a pregnancy within the next year;
18. Known to have, or suspected, allergy to materials contained in ORBERA™;
19. Participation in previous (within 60 days of study day 1) or ongoing clinical trial or current or past usage (within 60 days of study day 1) of investigational drug or device, or any use of an intragastric balloon prior to this study;
20. Genetically caused obesity;
21. Prior bariatric surgery or considering bariatric surgery during the study ;
22. Concomitant use of, or unwillingness to avoid any use of, weight loss medications, weight loss supplements, or weight loss herbal preparations;
23. Has a condition or is in a situation which in the Investigator's opinion may put the subject at significant risk or may interfere significantly with the subject's participation in the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese adults (22 years of age and older) with a Body Mass Index (BMI) of ≥ 30 kg/m2 and BMI ≤ 40 kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events (SAEs) | 26 weeks
  Incidence of device and procedure-related Serious Adverse Events (SAEs) after 26 weeks of ORBERA™ treatment will be no greater than 15%

SECONDARY OUTCOMES:
Percentage of Total Body Weight Loss (%TBWL) | 26 weeks
  To demonstrate that the mean percent Total Body Weight Loss (%TBWL) will be greater than 7.5% at ORBERA™ treatment conclusion (study week 26)
Adverse Events (AEs) | 12 months
  To continuously assess the safety of ORBERA™ by summarizing the occurrence of device- and procedure-related Adverse Events (AEs)
Serious Adverse Events (SAEs) | 12 months
  To continuously assess the safety of ORBERA™ by summarizing the occurrence of the following device- or procedure-related SAEs: gastric ulcers, esophageal injury, placement and removal related SAEs, early device removals, and balloon deflations
Total Body Weight Loss (%TBWL) | 12 months
  To estimate the %TBWL at each time point
Percentage of Excess Weight Loss (%EWL) | 12 months
  To estimate the percent Excess Weight Loss (%EWL) at each time point, assuming an ideal weight based on having a BMI of 25 kg/m2
Body Mass Index | 12 months
  To estimate the change from baseline in BMI at each time point
Nutritional Appetite Questionnaire | 12 months
  Will collect data on appetite, feelings of fullness, taste, and eating habits through a patient questionnaire.
Subject Treatment Satisfaction Survey | 12 months
  The Subject Satisfaction Survey will collect data on the subject's level of satisfaction with ORBERA treatment and their recommendation of ORBERA™ treatment to others.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L. Naveira, Study Director — Apollo Endosurgery, Inc.; James M Buswold, Study Director — Apollo Endosurgery, Inc.
Locations (11):
- United States (11):
  - Applied Research Center of Arkansas, Inc, Little Rock, Arkansas
  - Ellner Bariatric, San Diego, California
  - Sun Coast Bariactrics, St. Petersburg, Florida
  - Metroeast Endoscopic Surgery Center, Fairview Heights, Illinois
  - Louisville Surgical Associates, Louisville, Kentucky
  - Digestive Health Center / Gastroroenterology Associates, Baton Rouge, Louisiana
  - Surgical Specialists of Louisiana, Metairie, Louisiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Allure Medical Spa, Mount Clemens, Michigan
  - Center for Metabolic and Bariatric Surgery, Cincinnati, Ohio
  - Dr. Keith's Wellness Options, Norman, Oklahoma

REFERENCES:
- [Derived] Moore RL, Eaton L, Ellner J. Safety and Effectiveness of an Intragastric Balloon as an Adjunct to Weight Reduction in a Post-Marketing Clinical Setting. Obes Surg. 2020 Nov;30(11):4267-4274. doi: 10.1007/s11695-020-04798-5. PMID 32617919